CLINICAL TRIAL: NCT04691479
Title: Adherence and Quality of Life of CPAP for Obstructive Sleep Apnea With an Intervention Based on Stratification and Personalization of Care Plans: a Randomized Controlled Trial
Brief Title: Adherence and Quality of Life of CPAP for Obstructive Sleep Apnea
Acronym: PIMA1-JO-PR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Healthcare Spain (Industry)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIMA1-3450; 3450 (Registry Identifier: Ethics Committee for Clinical Research)
Record Dates: First submitted 2020-12-21; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: CPAP; Sleep Apnea; Adherence; Quality of Life
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Masking Description: After confirming their participation in the study, the patient was randomly assigned to one group or another, receiving the treatment as established in the protocol according to group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIMAGroup (Experimental): 1. Educational and training program using motivational interview technical.
  2. Stratification labels: to determine the personalized intervention plan are obtained from two types of variables: personal and modulation variables. For psychological variables the Perceived Competence Evaluation Questionnaire validated in Adherence to CPAP in OSA (CEPCA) is used. Drowsiness is obtained through the administration of the Epworth Somnolence Test, and the apnoea-hypopnea index is taken from the patient's clinical history.
  3. Segmentation: With the psychological and clinical variables, in this first visit, "predictive" information is obtained on how the patient's adherence will be: high adherence, moderate adherence or low adherence.
  4. Taking this information into account, the care plan will start considering how the patient is and their situation with respect to adherence. Depending on their evolution, the care plan is adapted. For patients with low adherence, telemonitoring is used.
  Interventions: Behavioral: Motivational Interview (MI) & Adherence Follow-Up
- Control (Experimental): The patients followed the standard of care, which consists of starting therapy in the hospital, where the nurse performed training in the use of CPAP equipment, mask adjustment, and safety and maintenance instructions. For follow-up, the patient was always referred to the Hospital, with a frequency established by the Spanish Society of Pulmonology and Thoracic Surgery (Day 30, Day 90 and Day 180). The follow-up procedure consisted of reviewing the CPAP hour meter and resolving any incidents that may have arisen, with the necessary corrective actions (change of mask, positive reinforcement, and explanation of specific aspects).
  Interventions: Behavioral: Adherence Follow-Up

INTERVENTIONS:
Behavioral: Motivational Interview (MI) & Adherence Follow-Up — 1. MEntA: Educational & Training Program
  2. Stratification: Identification of Personal Variables (Age, Level of study, Work status, preference of care attention, digital behaviour)
  3. Adherence evaluation: Evaluation of Perceived Competence, Quality of Life, Mood, Activities, Social relations and Social Support
  4. Identification of Care plan and Schedule next visits
  5. Follow-up D30-D60-D90-D180 depending of the care plan, through the channel that belong for each care plan
  Arms: PIMAGroup
Behavioral: Adherence Follow-Up — The nurse takes the compliance of the CPAP device, and ask to the patient if he had some problems.
  Arms: Control

SUMMARY:
A multicentre, randomized controlled trial (RCT) design.The control group followed the usual treatment, while the intervention group (PIMA) followed the treatment with an adapted and flexible care plan depending on socio-demographic, clinical and psychological variables. The treatment plan includes different channels (home, telephone, care center), a continuous evaluation, and the use of the motivational interview in each of the interventions with the patient. The main outcome was adherence. Secondary outcomes were quality of life, emotional state, activities, social relationships, perceived competence and motivation.

DETAILED DESCRIPTION:
The aim of this trial was to determine adherence to CPAP and health- related outcomes in patients with OSA via a comprehensive and multidisciplinary program based on stratification and individualized care plans, including the motivational interview.

A multicentre, randomized controlled trial (RCT) design was used. The control group followed the usual treatment, while the intervention group (PIMA) followed the treatment with an adapted and flexible care plan depending on socio-demographic, clinical and psychological variables. The treatment plan includes different channels (home, telephone, care center), a continuous evaluation, and the use of the motivational interview in each of the interventions with the patient. The main outcome was adherence. Secondary outcomes were quality of life, emotional state, activities, social relationships, perceived competence and motivation.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Diagnosis of OSA confirmed by sleep studies with polygraphy (PS) and / or polysomnography (PSG)

Exclusion Criteria:

* Subjects with obesity-related hypoventilation
* Severe COPD (chronic obstructive pulmonary disease)
* Cognitive disorders and those unable to understand the consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Adherence (changes) | Day 90, Day 180
  Number of hours of use of CPAP per night
Somnolence (changes) | Day 1, Day 90, Day 180
  Residual sleepiness after use of CPAP. Epworth Sleepiness Scale. Minimum score: 0; Maximum: 24. Higher scores=worse outcome
Perceived Competence (changes) | Day 1, Day 90, Day 180
  Self-Efficacy in the CPAP treatment. Perceived Competence Evaluation Questionnaire. Minimum score: 0; Maximum score 13. Higher score= Better outcome.

SECONDARY OUTCOMES:
Quality of Life (Changes) | Day 1, Day 90, Day 180
  Well-Being of the patient related to sleep apnea. Analogical Well-Being in Sleep Apnea Scale. Mininum score: 0; Maximum score: 10. Higher score= better outcome.
Mood (Changes) | Day 1, Day 90, Day 180
  Emotional status related to sleep apnea. Ad hoc question. Minimum score: 0; maximum score: 3. Higher score: Better outcome.
Activities (Changes) | Day 1, Day 90, Day 180
  Improving general activity after use CPAP. Ad hoc question. Minimum score: 0; maximum score: 3. Higher score: Better outcome.
Social Relations (Changes) | Day 1, Day 90, Day 180
  Improving general social relations after use CPAP. Ad hoc question. Minimum score: 0; maximum score: 3. Higher score: Better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Landete, PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- David Rudilla, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publication of results in two phases:
  * National Congress in Portugal
  * Publication in Research Journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the moment we are presenting the results in a journal for publication. The data may be requested from any of the researchers, and may be consulted online, the data being 100% anomized. Data accessibility will be in the next 36 months after publication.
Access Criteria: Researchers and reviewers

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT04691479/Prot_SAP_ICF_000.pdf